CLINICAL TRIAL: NCT01312922
Title: Pipamperone/Citalopram (PNB01) Versus Citalopram (CIT) and Versus Pipamperone (PIP) in the Treatment of Moderate to Severe Major Depressive Disorder (MDD): a Randomized, Double-blind Phase III Study of 10 Weeks
Brief Title: Pipamperone/Citalopram (PNB01) Versus Citalopram (CIT) and Versus Pipamperone (PIP) in Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaNeuroBoost N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNB01-C301; 2011-001190-11 (EudraCT Number)
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram; pipamperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PNB01 (Experimental): oral, once daily administration
  Interventions: Drug: PNB01 fixed dose combination of pipamperone and citalopram
- citalopram (Active Comparator): oral, once daily administration
  Interventions: Drug: Citalopram
- pipamperone (Sham Comparator): oral, once daily administration
  Interventions: Drug: Pipamperone

INTERVENTIONS:
Drug: PNB01 fixed dose combination of pipamperone and citalopram — oral once daily administration
  Arms: PNB01
Drug: Citalopram — oral once daily administration
  Arms: citalopram
Drug: Pipamperone — oral once daily administration
  Arms: pipamperone

SUMMARY:
The overall objective of this trial is to demonstrate clinically relevant superior antidepressant efficacy of the fixed dose combination PNB01 (low dose pipamperone and citalopram) over reference antidepressant treatment with citalopram alone, and a low dose of psychoactive pipamperone alone in patients with moderate to severe Major Depressive Disorder.

This study was specifically designed to assess patient related outcome (PRO) parameters using an Interactive Voice Response System (IVRS) via telephone.

DETAILED DESCRIPTION:
This is an international, double-blind, centrally randomized (stratified), multicenter study in 555 patients suffering from moderate to severe MDD in up to 40 sites in the USA, Germany and Canada. Eligible out-patients will be treated once daily (QD) with a fixed dose of either PNB01 (PIP 15 mg / CIT 20 mg (Week 1) - PIP 15 mg / CIT 40 mg (Week 2-10)), CIT alone (CIT 20 mg (Week 1) - CIT 40 mg (Week 2-10) or PIP 15 mg alone (Week 1-10) in a 1:1:1 ratio in a double-blind fashion for 10 weeks. Study visits will be conducted 1, 2, 3, 4, 6, 8 and 10 weeks after study treatment initiation. Possible withdrawal effects will be assessed 1 week after study treatment withdrawal.

A blood sample for pharmacokinetic analysis will be collected when drawing blood for routine biochemistry. Patients who provided written informed consent to participate to the study will be asked to provide their consent to participate also to the non-mandatory pharmacogenetic study.

Patient related outcomes will be collected electronically (ePRO) at study visits prior to visiting the investigator by using an Interactive Voice Response System (IVRS) via telephone. Patients wishing or choosing to discontinue the study treatment prematurely will be encouraged to continue to provide their scores, safety data and medications taken, up to the scheduled study end, by telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent.
2. Patient understands the investigational nature of the trial and is willing and able to comply with the trial requirements.
3. Patient is male or female, aged ≥ 18 years.
4. Patient has MDD according to the DSM IV-R criteria with an existence of depressed mood (DSM-IV-R Crit. A1) and loss of interest/anhedonia (DSM-IV-R Crit. A2) as confirmed by the MINI, lasting for at least 4 weeks and no longer than 18 months (78 weeks) for the current episode, and causing significant functional impairment (DSM-IV-R MDD C- criterion).
5. CGI-S rating of at least 4 and a minimum MADRS total score of 26 using IVRS ePRO at Baseline.

Exclusion Criteria:

1. Patient is pregnant, nursing, or is a woman of child-bearing potential who is not surgically sterile, 2 years postmenopausal, or who does not consistently use 2 combined effective methods of contraception (including at least 1 barrier method), unless sexually abstinent.
2. Existence of Mood Disorder with psychotic features and/or high suicidality risk, as confirmed by MINI.
3. Concomitant diagnosis of any additional primary Axis I disorder and presence of any of the following co-morbid disorders: (Hypo)manic episode, Panic Disorder (limited symptom attacks allowed), Obsessive Compulsive Disorder, Post-traumatic Stress Disorder, Alcohol dependence, any other Substance abuse and/or dependence, Psychotic Disorder, Eating Disorder, or General Anxiety Disorder, as confirmed by MINI.
4. Concomitant diagnosis of any primary Axis II disorder.
5. Patient is hospitalized.
6. Patient has a clinically relevant renal dysfunction (e.g. GFR <60mL/min).
7. Patient has hepatic dysfunction (total bilirubin >2.0mg/dL or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than 2 times the upper limit of the reference range).
8. Patient has a malignant neoplastic disease, a documented history of epilepsy (juvenile convulsions excepted) or a documented, in the opinion of the investigator, clinically relevant risk of bleeding (eg. severe bleeding disorder, treatment with warfarin, …).
9. Patient with a documented history or concomitant diagnosis or significant risk of cardiac arrhythmia or dysrhythmia, including a QTc interval of ≥500 ms at Baseline.
10. Patient has any other medical or psychiatric condition, which in the opinion of the investigator, can jeopardize or would compromise the patient's ability to participate in this trial or that would interfere with trial assessments.
11. Patient with documented alcohol or drug abuse, or having a positive standard screen for alcohol or drugs (including benzodiazepines and opioids).
12. Patient received, in the past 7 days treatment with any psychoactive drug prior to randomization, including typical and atypical antipsychotics, hypnotics, antidepressants, anxiolytic drugs, anticonvulsive therapy, opioids, monoamine oxidase (MAO) inhibitors, sedative antihistamines, psychostimulants or amphetamines, dopamine D2 receptor antagonists, butyrophenones, metoclopramide, lithium, anticonvulsants, benzodiazepines, or barbiturates. If patient has received such therapy, a washout period of at least 7 days prior to baseline is required before inclusion in this trial (except fluoxetine: 4 weeks, and St John's Wort or MAO inhibitors: within 2 weeks).
13. Concomitant treatment with diuretics, QT prolongation drugs, or dopamine agonists.
14. Resistant depression defined as having failed to respond to either: a/ 2 previous antidepressants at an adequate dose administered for at least 4 weeks during the current episode; b/ augmentation therapy with any atypical antipsychotic drug
15. Electroconvulsive therapy (ECT) or repetitive Transcranial Magnetic Stimulation therapy (rTMS) within the last 6 months; Vagus Nerve Stimulation (VNS) or Deep Brain Stimulation (DBS) ever.
16. Formal psychotherapy or alternative treatment for 1 week prior to or during the study.
17. Patient has participated in another trial of an investigational agent (including medical device) within the last 3 months prior to baseline or is currently participating in another trial of an investigational drug.
18. Known hypersensitivity to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Thase, MD, Study Chair — Director, Mood and Anxiety Section; 3535 Market Street, Suite 670; Philadelphia, PA 19104-3309, United States of America; Max Schmauss, MD, Study Chair — Bezirkskrankenhaus Augsburg Klinik für Psychiatrie, Psychotherapie und Psychosomatik Dr.-Mack-Straße 1 D-86156 Augsburg, Germany; Philippe Lemmens, PhD, Study Director — Pharmaneuroboost N.V. Alkerstraat 30A B-3570 Alken, Belgium
Locations (31):
- United States (26):
  - Site 103, Glendale, California
  - Site 101, National City, California
  - Site 113, Riverside, California
  - Site 106, San Diego, California
  - Site 116, San Diego, California
  - Site 112, Fort Myers, Florida
  - Site 135, Miami, Florida
  - Site 108, Winter Park, Florida
  - Site 133, Atlanta, Georgia
  - Site 128, Smyrna, Georgia
  - Site 132, Libertyville, Illinois
  - Site 117, Schaumburg, Illinois
  - Site 110, Baltimore, Maryland
  - Site 109, Flowood, Mississippi
  - Site 115, New York, New York
  - Site 126, Beachwood, Ohio
  - Site 127, Cincinnati, Ohio
  - Site 124, Middleburg Heights, Ohio
  - Site 105, Allentown, Pennsylvania
  - Site 123, Media, Pennsylvania
  - Site 122, Philadelphia, Pennsylvania
  - Site 119, Austin, Texas
  - Site 104, Dallas, Texas
  - Site 102, Wichita Falls, Texas
  - Site 107, Kirkland, Washington
  - Site 134, Seattle, Washington
- Canada (5):
  - Site 201, Kelowna, British Columbia
  - Site 202, Penticton, British Columbia
  - Site 205, Chatham, Ontario
  - Site 203, Mississauga, Ontario
  - Site 204, Mississauga, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a centrally randomized (stratified), double-blind, multicenter study in up to 40 sites in the U.S. and Canada.
Pre-assignment Details: A total of 555 eligible patients were planned and randomized in the study
Period: Overall Study
Arm/Group | PNB01 | Citalopram | Pipamperone
Started | 185 | 185 | 185
Completed | 117 | 131 | 135
Not Completed | 68 | 54 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PNB01 | Citalopram | Pipamperone | Total
Number analyzed (Participants) | 185 | 185 | 185 | 555
Age, Customized [Count of Participants; unit: Participants]
  18 - 60 years | 184 | 182 | 179 | 545
  > 60 years | 1 | 3 | 6 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 104 | 114 | 329
  Male | 74 | 81 | 71 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 1 | 7
  Asian | 5 | 6 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 53 | 54 | 54 | 161
  White | 116 | 119 | 120 | 355
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Early and Sustained (Antidepressant) Response (ESR) Rate
Description: Early and Sustained Response (ESR) is defined as a MADRS total score reduction from Baseline of 50% or more and a MADRS total score ≤16 at Week 2, Week 3, Week 4, and Week 6.
Time Frame: From (end of) Week 2 visit to (end of) Week 6 visit
Population: Full Analysis Set (FAS): The FAS consists of all patients who are randomized and were administered at least one dose of trial medication, as assessed from pill counting. Patients will be analyzed according to the treatment group to which they were randomized (intention-to-treat principle), irrespective of the study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | PNB01 | Citalopram | Pipamperone
Number analyzed (Participants) | 176 | 174 | 181
Participants | 17 | 17 | 17
Statistical Analysis 1: Comparison: PNB01 vs Citalopram; Test type: Superiority; p = 1.000, Fisher Exact; Odds Ratio (OR) = 0.987, 95% CI 2-sided [0.456 to 2.140]
Statistical Analysis 2: Comparison: PNB01 vs Pipamperone; Test type: Superiority; p = 1.000, Fisher Exact; Odds Ratio (OR) = 1.031, 95% CI 2-sided [0.476 to 2.233]

2. Secondary Outcome: Change From Baseline in Total MADRS Score at Week 6
Description: Change from baseline in total score on the Montgomery-Asberg Depression Rating Scale (MADRS) after 6 weeks of study treatment as assessed by the patient using an Interactive Voice Response System (IVRS) via telephone
  The MADRS scale is a widely used and well-validated 10-item diagnostic questionnaire designed to measure the severity of depressive episodes in patients with mood disorders. The 10 items are all rated on a scale from 0 to 6 (resulting in a maximum total score of 60 points) and include 'apparent sadness', 'reported sadness', 'inner tension', 'reduced sleep', 'reduced appetite', 'concentration difficulties', 'lassitude', 'inability to feel', 'pessimistic thoughts' and 'suicidal thoughts'. Higher scores indicative of greater depressive symptomology.
Time Frame: From Baseline (Day 1) to (end of) Week 6
Population: Secondary Outcome Measures were pre-specified to be completed based on significance of the Primary Outcome Measure. Secondary Outcome Measures were therefore not completed.
Arm/Group | PNB01 | Citalopram | Pipamperone
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Total SDS Score at Week 6
Description: Change from baseline in total score on the Sheehan Disability Scale (SDS) after 6 weeks of study treatment as assessed by the patient using an Interactive Voice Response System (IVRS) via telephone
  The SDS is a generic brief self-report tool that was developed to assess functional impairment in three inter-related domains; 1) work or school, 2) social life and 3) family life. The patient rates the extent to which work/school, social life and home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale. Total scores range from a minimum of 0 to a maximum of 30 (0 unimpaired, 30 highly impaired).
Time Frame: From Baseline (Day 1) to (end of) Week 6 visit
Population: as for outcome 2
Arm/Group | PNB01 | Citalopram | Pipamperone
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks + follow-up 1 week
Description: Safety Set (SS): The SS consists of all patients who are randomized and were administered at least 1 dose of trial medication, as assessed from pill counting. Patients will be analyzed according to the treatment group of the study treatment that was actually received.
Arm/Group | PNB01 | Citalopram | Pipamperone
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/185 | 0/185
Serious Adverse Events (participants affected / at risk) | 3/185 | 4/185 | 1/185
Other Adverse Events (participants affected / at risk) | 127/185 | 131/185 | 118/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNB01 (N=185) | Citalopram (N=185) | Pipamperone (N=185)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
dehydratation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNB01 (N=185) | Citalopram (N=185) | Pipamperone (N=185)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 17 (19) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 18 (18) | 10 (11) | 16 (17)
Nausea (Gastrointestinal disorders) | 16 (17) | 28 (30) | 14 (16)
Dizziness (Nervous system disorders) | 10 (13) | 12 (14) | 10 (11)
Headache (Nervous system disorders) | 20 (20) | 20 (25) | 19 (21)
Sedation (Nervous system disorders) | 4 (5) | 7 (7) | 8 (8)
Somnolence (Nervous system disorders) | 29 (29) | 20 (23) | 12 (13)
Insomnia (Psychiatric disorders) | 11 (12) | 20 (20) | 9 (10)
Fatigue (General disorders) | 6 (7) | 9 (10) | 5 (6)
Nasopharyngitis (Infections and infestations) | 8 (8) | 10 (10) | 6 (6)
Weight Increase (Investigations) | 9 (10) | 2 (2) | 15 (15)
Decreased Appetitie (Metabolism and nutrition disorders) | 4 (5) | 10 (11) | 3 (3)

LIMITATIONS AND CAVEATS:
To avoid limited risk of concluding efficacy when there is no effect, hierarchical testing was implemented with following order of confirmatory tests: 1) Patient-ESR rates of PNB01vs citalopram 2) If above testing is sig., repeat patient-ESR testing for PNB01vs pipamperone 3) In case in 1 of these 2 tests PNB01 does not have sig. higher ESR rate, trial is considered negative, & no following sec. confirmatory tests are to be executed.

Secondary Outcome Measures were therefore not completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No